CLINICAL TRIAL: NCT01369537
Title: Neurological Impact of Vascular Events In Noncardiac Surgery patIents cOhort evaluatioN Pilot Study
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: NeuroVISION Pilot
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Perioperative Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- adults > 65 yrs undergoing noncardiac surgery

SUMMARY:
Two hundred million adults worldwide have major surgery every year. A million of these patients will have an obvious stroke after their surgery. Another 10 million patients may have "silent" strokes. Although silent strokes are not diagnosed immediately, they are likely to reduce patients' short-term memory, concentration, and ability to function at home. However, the investigators do not know how common silent strokes are after noncardiac surgery, nor the extent to which they affect brain function.

The investigators will first perform a pilot trial to determine the feasibility of the larger study that will provide the definitive answer to this question. Participating patients will be assessed by questionnaire before and after surgery, and will have a magnetic resonance imaging (MRI) study of the brain after the surgery to look for silent strokes. Combining the results of the MRI and the questionnaires will allow us to determine the frequency of silent strokes after non-cardiac surgery, and their effect on brain function. The NeuroVISION Pilot Study will determine the feasibility of a large study to examine the frequency and the impact of silent stroke in patients who undergo noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 65,
* undergoing noncardiac surgery,
* regional or general anesthetic.

Exclusion Criteria:

-Patients who have a contraindication to MRI.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years and older undergoing noncardiac surgery and staying in hospital overnight.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: PJ Devereaux, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Mrkobrada M, Hill MD, Chan MT, Sigamani A, Cowan D, Kurz A, Sessler DI, Jacka M, Graham M, Dasgupta M, Dunlop V, Emery DJ, Gulka I, Guyatt G, Heels-Ansdell D, Murkin J, Pettit S, Sahlas DJ, Sharma M, Sharma M, Srinathan S, St John P, Tsai S, Gelb AW, O'Donnell M, Siu D, Chiu PW, Sharath V, George A, Devereaux PJ. Covert stroke after non-cardiac surgery: a prospective cohort study. Br J Anaesth. 2016 Aug;117(2):191-7. doi: 10.1093/bja/aew179. PMID 27440630